CLINICAL TRIAL: NCT06950216
Title: Intraoperative Neuromonitoring During Radical Prostatectomy
Brief Title: IONM During Radical Prostatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: KY-2025-007
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Intraoperative neuromonitoring; Urinary incontinence; Erectile dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IONM group (Experimental): IONM was performed during the operation.
  Interventions: Other: IONM
- control group (No Intervention): No IONM

INTERVENTIONS:
Other: IONM — The probe needle electrodes were inserted into the corpus cavernosum penis, ischiocavernosus muscle, bulbocavernosus muscle, anal sphincter, etc., and each monitoring electrode was connected to the nerve monitor. The changes of electromyography of each effector during the operation were monitored in real time. The stimulation electrode was placed in the abdominal cavity during the operation. During the resection of the prostate, electrical stimulation was performed on the possible running area of the NVB, and the stimulation site where the signal was monitored was protected from resection and burning under the premise of safe surgery.
  Arms: IONM group

SUMMARY:
At present, the preferred treatment for patients with prostate cancer is still radical prostatectomy. Postoperative patients often face some complications, the most common complications include urinary incontinence and erectile dysfunction. Urinary incontinence is caused by intraoperative injury of urinary control nerves or muscles. Erectile dysfunction is related to intraoperative injury of nerves that control erection. Therefore, intraoperative nerve preservation is a key measure to reduce postoperative complications, especially to prevent erectile dysfunction. This study intends to improve the nerve-sparing radical prostatectomy by monitoring the nerve during radical prostatectomy, locating the cavernous nerve and other related nerves, in order to reduce the incidence of postoperative complications such as erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

- 1: Prostate cancer patients undergoing surgical treatment in our Hospital 2: Understand the content of this study, actively provide complete and true medical history and examination data, and be willing to cooperate with postoperative interviewers.

3: Voluntarily participate in the study and sign the treatment document within the ethical framework.

Exclusion Criteria:

* 1: Histopathology showed that the patient did not have prostate cancer 2: Use a cardiac pacemaker or other electromechanical prosthesis device 3: Suffering from a serious neurological disease, mental illness or other illness that may be life-threatening within two years

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 | 1,3,6 and 12 months after operation
  international index of erectile function-5

CONTACTS AND LOCATIONS:
Overall Officials: Yichun Zheng, Doctor, Study Chair — The Fourth Affiliated Hospital Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No